CLINICAL TRIAL: NCT02713204
Title: A Randomized, Double-Masked, Active-Controlled Phase 2 Study of the Efficacy, Safety, and Tolerability of Repeated Doses of Intravitreal REGN910-3 in Patients With Neovascular Age-Related Macular Degeneration
Brief Title: Anti-angiOpoeitin 2 Plus Anti-vascular eNdothelial Growth Factor as a therapY for Neovascular Age Related Macular Degeneration: Evaluation of a fiXed Combination Intravitreal Injection
Acronym: ONYX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R910-3-AMD-1517
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Neovascular Age-Related Macular Degeneration
MeSH Terms: interventions — aflibercept; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- REGN910-3 (3 mg: 2 mg) (Experimental): Participants were administered intravitreal injection of REGN910-3 (3 milligram [mg]:2 mg) every 4 weeks (Q4) on Day 1, Week 4, and Week 8 for 3 initial doses followed by every Week 8 (Q8) dosing beginning at Week 16 up to Week 32.
  Interventions: Drug: REGN910-3
- REGN910-3 (6 mg:2 mg) (Experimental): Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses. At Week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) Q8 or Q12 (beginning at Week 16 or Week 20) through Week 32.
  Interventions: Drug: REGN910-3
- Aflibercept (IAI) 2 mg (Experimental): Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q8 or Q12 (beginning at Week 16 or 20) or REGN910-3 (6 mg:2 mg) Q8 beginning at Week 16 through Week 32.
  Interventions: Drug: REGN910-3; Drug: Intravitreal Aflibercept Injection (IAI)

INTERVENTIONS:
Drug: REGN910-3
Drug: Intravitreal Aflibercept Injection (IAI)
  Other Names: EYLEA® (aflibercept) Injection; BAY86-5321
  Arms: Aflibercept (IAI) 2 mg

SUMMARY:
The primary objective of the study is to compare the efficacy of intravitreal (IVT)-administered REGN910-3 compared to intravitreal aflibercept injection (IAI).

ELIGIBILITY:
Key Inclusion Criteria:

1. Men or women ≥50 years of age with active subfoveal CNV secondary to AMD, including juxtafoveal lesions that affect the fovea as evidenced by FA in the study eye as assessed by a central reading center
2. BCVA ETDRS letter score of 73 to 24 (Snellen equivalent of 20/40 to 20/320) in the study eye.
3. Willing and able to comply with clinic visits and study-related procedures.
4. Provide signed informed consent.

Key Exclusion Criteria:

1. Evidence of CNV due to any cause other than AMD in either eye
2. Prior IVT anti-VEGF in the study eye
3. Evidence of DME or diabetic retinopathy (defined as more than 1 microaneurysm) in either eye in diabetic patients
4. Any history of macular hole of stage 2 and above in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (87):
- United States (87):
  - Regeneron Investigational Site, Mobile, Alabama
  - Regeneron Investigational Site 1, Phoenix, Arizona
  - Regeneron Investigational Site 2, Phoenix, Arizona
  - Regeneron Investigational Site 3, Phoenix, Arizona
  - Regeneron Investigational Site 1, Tucson, Arizona
  - Regeneron Investigational Site 2, Tucson, Arizona
  - Regeneron Investigational Site, Arcadia, California
  - Regeneron Investigational Site, Bakersfield, California
  - Regeneron Investigational Site, Beverly Hills, California
  - Regeneron Investigational Site, Encino, California
  - Regeneron Investigational Site 1, Los Angeles, California
  - Regeneron Investigational Site 2, Los Angeles, California
  - Regeneron Investigational Site, Mountain View, California
  - Regeneron Investigational Site, Oceanside, California
  - Regeneron Investigational Site 1, Palm Desert, California
  - Regeneron Investigational Site 2, Palm Desert, California
  - Regeneron Investigational Site, Palo Alto, California
  - Regeneron Investigational Site, Poway, California
  - Regeneron Investigational Site, Redlands, California
  - Regeneron Investigational Site, Sacramento, California
  - Regeneron Investigational Site, Santa Maria, California
  - Regeneron Investigational Site, New London, Connecticut
  - Regeneron Investigational Site, Altamonte Springs, Florida
  - Regeneron Investigational Site, Fort Lauderdale, Florida
  - Regeneron Investigational Site, Lakeland, Florida
  - Regeneron Investigational Site, Largo, Florida
  - Regeneron Investigational Site, Miami, Florida
  - Regeneron Investigational Site, Naples, Florida
  - Regeneron Investigational Site, Palm Beach, Florida
  - Regeneron Investigational Site, Tallahassee, Florida
  - Regeneron Investigational Site, Winter Haven, Florida
  - Regeneron Investigational Site, Augusta, Georgia
  - Regeneron Investigational Site, Decatur, Georgia
  - Regeneron Investigational Site, ‘Aiea, Hawaii
  - Regeneron Investigational Site 1, Chicago, Illinois
  - Regeneron Investigational Site 2, Chicago, Illinois
  - Regeneron Investigational Site, Lemont, Illinois
  - Regeneron Investigational Site, Oak Forest, Illinois
  - Regeneron Investigational Site, Oak Park, Illinois
  - Regeneron Investigational Site, Urbana, Illinois
  - Regeneron Investigational Site, New Albany, Indiana
  - Regeneron Investigational Site, Des Moines, Iowa
  - Regeneron Investigational Site, Metairie, Louisiana
  - Regeneron Investigational Site 1, Baltimore, Maryland
  - Regeneron Investigational Site 2, Baltimore, Maryland
  - Regeneron Investigational Site, Chevy Chase, Maryland
  - Regeneron Investigational Site 1, Boston, Massachusetts
  - Regeneron Investigational Site 2, Boston, Massachusetts
  - Regeneron Investigational Site, Jackson, Michigan
  - Regeneron Investigational Site, Minneapolis, Minnesota
  - Regeneron Investigational Site, St Louis, Missouri
  - Regeneron Investigational Site, Las Vegas, Nevada
  - Regeneron Investigational Site, Portsmouth, New Hampshire
  - Regeneron Investigational Site, Edison, New Jersey
  - Regeneron Investigational Site, Teaneck, New Jersey
  - Regeneron Investigational Site, Albuquerque, New Mexico
  - Regeneron Investigational Site, Albany, New York
  - Regeneron Investigational Site, Bloomfield, New York
  - Regeneron Investigational Site, Great Neck, New York
  - Regeneron Investigational Site, Hauppauge, New York
  - Regeneron Investigational Site, Rochester, New York
  - Regeneron Investigational Site, Syracuse, New York
  - Regeneron Investigational Site, Asheville, North Carolina
  - Regeneron Investigational Site, Charlotte, North Carolina
  - Regeneron Investigational Site, Durham, North Carolina
  - Regeneron Investigational Site, Cleveland, Ohio
  - Regeneron Investigational Site, Dublin, Ohio
  - Regeneron Investigational Site, Portland, Oregon
  - Regeneron Investigational Site, Camp Hill, Pennsylvania
  - Regeneron Investigational Site, Huntingdon, Pennsylvania
  - Regeneron Investigational Site, Ladson, South Carolina
  - Regeneron Investigational Site, Rapid City, South Dakota
  - Regeneron Investigational Site, Germantown, Tennessee
  - Regeneron Investigational Site, Knoxville, Tennessee
  - Regeneron Investigational Site, Nashville, Tennessee
  - Regeneron Investigational Site, Abilene, Texas
  - Regeneron Investigational Site 1, Austin, Texas
  - Regeneron Investigational Site 2, Austin, Texas
  - Regeneron Investigational Site, Dallas, Texas
  - Regeneron Investigational Site 1, Fort Worth, Texas
  - Regeneron Investigational Site 2, Fort Worth, Texas
  - Regeneron Investigational Site, Harlingen, Texas
  - Regeneron Investigational Site, Houston, Texas
  - Regeneron Investigational Site, The Woodlands, Texas
  - Regeneron Investigational Site, Willow Park, Texas
  - Regeneron Investigational Site, Salt Lake City, Utah
  - Regeneron Investigational Site, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 87 sites in the United States. A total of 560 participants were screened in the study.
Pre-assignment Details: Out of 560 participants, 365 were randomized & treated. Participants were randomized in 1:2:3 to receive REGN910-3 3:2mg, REGN910-3 6:2mg & 2mg intravitreal aflibercept injection (IAI) followed by re-randomization at week 12 in REGN910-3 6:2mg & IAI 2mg arm. Not all participants who completed Week 12 were re-randomized & continued to Week 36.
Groups:
- REGN910-3 (3 mg:2 mg): Participants were administered intravitreal injection of REGN910-3 (3 milligram [mg]:2 mg) every 4 weeks (Q4) on Day 1, Week 4, and Week 8 for 3 initial doses followed by every Week 8 (Q8) dosing beginning at Week 16 through Week 32.
- Aflibercept 2 mg: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q8 or Q12 (beginning at Week 16 or 20) or REGN910-3 (6 mg:2 mg) Q8 beginning at Week 16 through Week 32.
- REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8: Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses. At Week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) Q8 beginning at Week 16 through Week 32.
- REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12: Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses. At week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) Q12 beginning at Week 20 through Week 32.
- Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At week 12, participants were re-randomized to receive IAI Q8 beginning at week 16 through week 32.
- Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q12 beginning at Week 20 through Week 32.
- Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) Q8 beginning at Week 16 through Week 32.
Period: Baseline (Day 1) up to Week 12
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 | Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Started | 60 | 122 | 183 | 0 | 0 | 0 | 0 | 0
Completed | 59 | 121 | 181 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: From Week 12 up to Week 36
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept 2 mg | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q8 | Aflibercept 2 mg Q4 to Aflibercept 2 mg Q12 | Aflibercept 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Started | 58 | 0 | 0 | 57 | 62 | 60 | 62 | 58
Completed | 57 | 0 | 0 | 53 | 60 | 59 | 60 | 54
Not Completed | 1 | 0 | 0 | 4 | 2 | 1 | 2 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Participant Re-located | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- REGN910-3 (3 mg:2 mg): Participants were administered intravitreal injection of REGN910-3 (3 mg:2 mg) every 4 weeks (Q4) on Day 1, Week 4, and Week 8 for 3 initial doses followed by every Week 8 (Q8) dosing beginning at Week 16 through Week 32.
- REGN910-3 (6 mg:2 mg): Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses. At Week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) at Week 16 or Week 20 and Q8 or Q12 through Week 32.
- Total: Total of all reporting groups
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept (IAI) 2 mg | Total
Number analyzed (Participants) | 59 | 122 | 183 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (9.37) | 79.4 (8.91) | 78.4 (8.37) | 78.9 (8.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 75 | 110 | 226
  Male | 18 | 47 | 73 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9 | 18
  Not Hispanic or Latino | 57 | 115 | 174 | 346
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 58 | 116 | 178 | 352
  Black or African American | 0 | 1 | 1 | 2
  Asian | 1 | 3 | 2 | 6
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Other | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 12
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. Best Corrected Visual Acuity (BCVA) score was measured using an eye chart and was reported as the number of letters read correctly at a testing distance of 4 meters using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. Change from baseline calculated by subtracting baseline value from observed post-baseline value at Week 12.
Time Frame: At Week 12
Population: Full analysis set included all randomized participants who received any study drug, had baseline measurement of BCVA & at least 1 post-baseline assessment of BCVA. Last observation carried forward (LOCF) method was used to impute missing data. Here "Overall Number of Participants Analyzed" = Participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Letters correctly read
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept (IAI) 2 mg
Number analyzed (Participants) | 59 | 122 | 183
Letters correctly read | 5.2 (10.51) | 5.6 (10.59) | 5.4 (9.85)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept (IAI) 2 mg; Test type: Superiority — Analysis was performed using analysis of covariance (ANCOVA) model with baseline measurement as a covariate and treatment group as fixed factors; p = 0.9894, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.02, 95% CI 2-sided [-2.99 to 3.03]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) vs Aflibercept (IAI) 2 mg; Analysis was performed using analysis of covariance (ANCOVA) model with baseline measurement as a covariate and treatment group as fixed factors; Test type: Superiority; p = 0.8346, ANCOVA; Least square mean difference = 0.25, 95% CI 2-sided [-2.09 to 2.59]

2. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Measured by Early Treatment Diabetic Retinopathy Study (ETDRS) Letter Score at Week 36
Description: Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at 4 meters. BCVA score was measured using an eye chart and was reported as the number of letters read correctly at a testing distance of 4 meters using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. Change from baseline calculated by subtracting baseline value from observed post-baseline value at Week 36.
Time Frame: At Week 36
Measure: Mean (Standard Deviation); unit: Letters correctly read
Groups:
- Aflibercept 2(IAI) mg Q4 to Aflibercept (IAI) 2 mg Q8: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q8 beginning at Week 16 through Week 32.
- Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q12 beginning at Week 20 through Week 32.
- Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) Q8 beginning at Week 16 through Week 32.
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept 2(IAI) mg Q4 to Aflibercept (IAI) 2 mg Q8 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12 | Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 58 | 57 | 62 | 60 | 62 | 58
Letters correctly read | 5.9 (11.95) | 6.0 (12.00) | 6.4 (12.24) | 6.9 (12.49) | 4.2 (12.50) | 2.9 (12.16)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept 2(IAI) mg Q4 to Aflibercept (IAI) 2 mg Q8; Analysis was performed using ANCOVA model with baseline measurement as a covariate, and treatment group and BCVA stratification variable as fixed factors; Test type: Superiority; p = 0.4611, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -1.20, 95% CI 2-sided [-4.41 to 2.00]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs Aflibercept 2(IAI) mg Q4 to Aflibercept (IAI) 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — Threshold for significance at 0.05 level; p = 0.2225, ANCOVA; Least square mean difference = -2.00, 95% CI 2-sided [-5.22 to 1.22]
Statistical Analysis 3: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept 2(IAI) mg Q4 to Aflibercept (IAI) 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6063, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.82, 95% CI 2-sided [-3.97 to 2.32]
Statistical Analysis 4: Comparison: Aflibercept 2(IAI) mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0426, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -3.25, 95% CI 2-sided [-6.39 to -0.11]
Statistical Analysis 5: Comparison: Aflibercept 2(IAI) mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0073, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -4.39, 95% CI 2-sided [-7.58 to -1.19]
Statistical Analysis 6: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4690, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 1.17, 95% CI 2-sided [-2.01 to 4.36]
Statistical Analysis 7: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1267, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 2.42, 95% CI 2-sided [-0.69 to 5.54]

3. Secondary Outcome: Change From Baseline in Central Sub-field Retinal Thickness (CST) Measured by Spectral Domain Optical Coherence Tomography (SD-OCT) at Week 12
Description: Central Sub-field Retinal Thickness (CST) was assessed using Spectral Domain Optical Coherence Tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from baseline indicated improvement. Change from baseline calculated by subtracting baseline value from last observation carried forward (LOCF) post-baseline value at Week 12.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept (IAI) 2 mg
Number analyzed (Participants) | 59 | 122 | 182
Microns | -182.2 (172.73) | -200.0 (152.82) | -178.6 (138.85)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept (IAI) 2 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.4130, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -11.57, 95% CI 2-sided [-39.5 to 16.20]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) vs Aflibercept (IAI) 2 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.6587, ANCOVA; Least square mean difference = -4.88, 95% CI 2-sided [-26.2 to 16.85]

4. Secondary Outcome: Change From Baseline in Central Sub-field Retinal Thickness (CST) Measured by Spectral Domain Optical Coherence Tomography (SD-OCT) at Week 36
Description: CST was assessed using spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. SD-OCT was performed in the study eye after pupil dilation. A negative change from baseline indicated improvement. Change from baseline calculated by subtracting baseline value from LOCF post-baseline value at Week 36.
Time Frame: At Week 36
Population: FAS secondary randomization set was used. Here "Overall Number of Participants Analyzed"= Participants who were evaluable for this endpoint.
Measure: Mean (Standard Deviation); unit: Microns
Groups:
- Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q8 beginning at Week 16 through Week 32.
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12 | Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 58 | 57 | 62 | 59 | 62 | 58
Microns | -174.6 (165.22) | -216.6 (187.40) | -181.3 (148.71) | -198.4 (155.72) | -169.7 (129.74) | -187.3 (161.72)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3833, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 17.04, 95% CI 2-sided [-21.35 to 55.43]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5141, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 12.85, 95% CI 2-sided [-25.84 to 51.53]
Statistical Analysis 3: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0785, ANCOVA; Least square mean difference = 33.89, 95% CI 2-sided [-3.89 to 71.67]
Statistical Analysis 4: Comparison: Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0281, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 42.27, 95% CI 2-sided [4.56 to 79.98]
Statistical Analysis 5: Comparison: Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; Test type: Superiority; p = 0.3934, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 16.65, 95% CI 2-sided [-21.67 to 54.96]
Statistical Analysis 6: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.2790, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 21.05, 95% CI 2-sided [-17.13 to 59.22]
Statistical Analysis 7: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6586, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -8.38, 95% CI 2-sided [-45.64 to 28.88]

5. Secondary Outcome: Change From Baseline in Choroidal Neovascularization (CNV) Area at Week 12
Description: Choroidal neovascularization (CNV) was evaluated using fluorescein angiography (FA).CNV area values measured in square millimeters (mm^2); lower values represent better outcomes.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept (IAI) 2 mg
Number analyzed (Participants) | 58 | 115 | 171
mm^2 | -2.2 (5.59) | -3.5 (5.34) | -3.7 (6.22)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept (IAI) 2 mg; Test type: Superiority; p = 0.4889, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.55, 95% CI 2-sided [-1.01 to 2.10]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) vs Aflibercept (IAI) 2 mg; Test type: Superiority; p = 0.7027, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.24, 95% CI 2-sided [-0.99 to 1.46]

6. Secondary Outcome: Change From Baseline in Choroidal Neovascularization (CNV) Area at Week 36
Description: as for outcome 5
Time Frame: At Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12 | Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 58 | 56 | 62 | 59 | 62 | 58
mm^2 | -3.7 (5.04) | -4.1 (6.09) | -4.9 (5.58) | -4.3 (6.55) | -5.1 (5.60) | -5.3 (5.19)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; Test type: Superiority; p = 0.4927, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.60, 95% CI 2-sided [-2.34 to 1.13]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; Test type: Superiority; p = 0.6645, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.38, 95% CI 2-sided [-1.36 to 2.13]
Statistical Analysis 3: Comparison: Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; Test type: Superiority; p = 0.3091, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.89, 95% CI 2-sided [-2.61 to 0.83]
Statistical Analysis 4: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; Test type: Superiority; p = 0.4898, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.60, 95% CI 2-sided [-2.29 to 1.10]
Statistical Analysis 5: Comparison: Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; Test type: Superiority; p = 0.3504, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.80, 95% CI 2-sided [-2.50 to 0.89]
Statistical Analysis 6: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; Test type: Superiority; p = 0.2632, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.98, 95% CI 2-sided [-2.70 to 0.74]
Statistical Analysis 7: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; Test type: Superiority; p = 0.8056, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.21, 95% CI 2-sided [-1.46 to 1.88]

7. Secondary Outcome: Change From Baseline in Total Lesion Area at Week 12
Description: Total lesion area was evaluated using fluorescein angiography (FA). Lesion area values measured in square millimeters (mm^2); lower values represent better outcomes.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept (IAI) 2 mg
Number analyzed (Participants) | 58 | 115 | 171
mm^2 | -2.0 (6.10) | -3.5 (5.45) | -3.4 (6.48)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept (IAI) 2 mg; Test type: Superiority; p = 0.5065, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.57, 95% CI 2-sided [-1.11 to 2.25]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) vs Aflibercept (IAI) 2 mg; Test type: Superiority; p = 0.7418, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.22, 95% CI 2-sided [-1.55 to 1.10]

8. Secondary Outcome: Change From Baseline in Total Lesion Area at Week 36
Description: as for outcome 7
Time Frame: At Week 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12 | Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 58 | 56 | 62 | 59 | 62 | 58
mm^2 | -3.0 (5.91) | -3.9 (5.79) | -4.7 (5.35) | -3.9 (6.67) | -4.7 (5.43) | -5.3 (5.20)
Statistical Analysis 1: Comparison: REGN910-3 (3 mg:2 mg) vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; Test type: Superiority; p = 0.8383, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.19, 95% CI 2-sided [-1.99 to 1.62]
Statistical Analysis 2: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; Test type: Superiority; p = 0.9180, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.10, 95% CI 2-sided [-1.91 to 1.72]
Statistical Analysis 3: Comparison: Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8; Test type: Superiority; p = 0.1238, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -1.41, 95% CI 2-sided [-3.20 to 0.39]
Statistical Analysis 4: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8; Test type: Superiority; p = 0.2819, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.97, 95% CI 2-sided [-2.73 to 0.80]
Statistical Analysis 5: Comparison: Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 vs Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; Test type: Superiority; p = 0.2581, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -1.02, 95% CI 2-sided [-2.78 to 0.75]
Statistical Analysis 6: Comparison: REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 vs REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12; Test type: Superiority; p = 0.3390, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = -0.87, 95% CI 2-sided [-2.66 to 0.92]
Statistical Analysis 7: Comparison: Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12; Test type: Superiority; p = 0.9558, ANCOVA — Threshold for significance at 0.05 level; Least square mean difference = 0.05, 95% CI 2-sided [-1.69 to 1.79]

9. Other Pre Specified Outcome: Proportion of Participants With No Retinal and/or Subretinal Fluid at Week 12
Description: Retinal and/or subretinal fluid was assessed using intraretinal fluid (IRF) cystoid edema and subretinal fluid (SRF) in the center subfield on optical coherence tomography (OCT). If answers were "no" to both measurements, there was no retinal and/or subretinal fluid (Dry); if "yes" to any of the 2 measurements, there was retinal and/or subretinal fluid (Not Dry); other than the previous 2 cases, retinal and/or subretinal fluid was undetermined.
Time Frame: At Week 12
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) | Aflibercept (IAI) 2 mg
Number analyzed (Participants) | 57 | 122 | 179
Proportion of participants | 0.49 | 0.51 | 0.44

10. Other Pre Specified Outcome: Proportion of Participants With No Retinal and/or Subretinal Fluid From Baseline Through Week 36
Description: Retinal and/or subretinal fluid was assessed using intraretinal fluid (IRF) cystoid edema and subretinal fluid (SRF) in the center subfield on OCT. If answers were "no" to both measurements, there was no retinal and/or subretinal fluid (Dry); if "yes" to any of the 2 measurements, there was retinal and/or subretinal fluid (Not Dry); other than the previous 2 cases, retinal and/or subretinal fluid was undetermined.
Time Frame: Baseline through Week 36
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12 | Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 57 | 57 | 62 | 59 | 62 | 55
Proportion of participants | 0.54 | 0.49 | 0.53 | 0.42 | 0.53 | 0.47

11. Other Pre Specified Outcome: Time to No Retinal and/or Subretinal Fluid Through Week 36
Description: Kaplan-Meier estimated time to no retinal and/or subretinal fluid through week 36 (days). Retinal and/or subretinal fluid was assessed using intraretinal fluid (IRF) cystoid edema and subretinal fluid (SRF). If answers were "no" to both measurements, there was no retinal and/or subretinal fluid (Dry); if "yes" to any of the 2 measurements, there was retinal and/or subretinal fluid (Not Dry); other than the previous 2 cases, retinal and/or subretinal fluid was undetermined.
Time Frame: Baseline through Week 36
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | REGN910-3 (3 mg:2 mg) | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q8 | REGN910-3 (6 mg:2 mg) Q4 to REGN910-3 (6 mg:2 mg) Q12 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q8 | Aflibercept (IAI) 2 mg Q4 to Aflibercept (IAI) 2 mg Q12 | Aflibercept (IAI) 2 mg Q4 to REGN910-3 (6 mg:2 mg) Q8
Number analyzed (Participants) | 58 | 57 | 62 | 60 | 62 | 58
Days | 105.6 (11.06) | 80.9 (9.02) | 84.9 (8.01) | 106.4 (11.04) | 96.5 (11.27) | 107.1 (10.05)

ADVERSE EVENTS:
Time Frame: Timeframe for AE reporting
Description: Reported adverse events are treatment-emergent adverse events that are AEs that developed/worsened during the study (Baseline through Week 36).
Groups:
- REGN910-3 3 mg:2 mg: Participants were administered intravitreal injection of REGN910-3 (3 mg:2 mg) every 4 weeks (Q4) on Day 1, Week 4, and Week 8 for 3 initial doses followed by every Week 8 (Q8) dosing beginning at Week 16 through Week 32.
- REGN910-3 6 mg:2 mg: Participants were administered intravitreal injection of REGN910-3 (6 mg:2 mg) Q4 on Day 1, Week 4 and Week 8 for 3 initial doses. At Week 12, participants were re-randomized to receive REGN910-3 (6 mg:2 mg) Q8 or Q12 (beginning at Week 16 or Week 20) through Week 32.
- IAI 2 mg: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q8 or Q12 (beginning at Week 16 or 20) or REGN910-3 (6 mg:2 mg) Q8 beginning at Week 16 through Week 32.
- IAI 2mg to REGN910-3: Participants were administered intravitreal injection of Aflibercept (IAI) 2 mg Q4 on Day 1, Week 4 and Week 8 for 3 initial doses up to Week 12. At Week 12, participants were re-randomized to receive IAI Q8 or Q12 (beginning at Week 16 or 20) or REGN910-3 (6 mg:2 mg) Q8 beginning at Week 16 through Week 32.
  Data in this arm include only the 58 participants that switched to high dose at week 16. Data from these 58 participants are also included in the Aflibercept (IAI) 2 mg arm (n = 183).
Arm/Group | REGN910-3 3 mg:2 mg | REGN910-3 6 mg:2 mg | IAI 2 mg | IAI 2mg to REGN910-3
All-Cause Mortality (participants affected / at risk) | 1/60 | 2/122 | 7/183 | 3/58
Serious Adverse Events (participants affected / at risk) | 11/60 | 20/122 | 30/183 | 8/58
Other Adverse Events (participants affected / at risk) | 17/60 | 41/122 | 51/183 | 20/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN910-3 3 mg:2 mg (N=60) | REGN910-3 6 mg:2 mg (N=122) | IAI 2 mg (N=183) | IAI 2mg to REGN910-3 (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardio-Respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (2) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REGN910-3 3 mg:2 mg (N=60) | REGN910-3 6 mg:2 mg (N=122) | IAI 2 mg (N=183) | IAI 2mg to REGN910-3 (N=58)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 4 (5) | 1 (2)
Dry eye (Eye disorders) | 2 (2) | 7 (8) | 4 (4) | 1 (1)
Neovascular age-related macular degeneration (Eye disorders) | 4 (4) | 5 (5) | 5 (5) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 2 (2) | 12 (14) | 6 (7)
Vitreous detachment (Eye disorders) | 3 (4) | 7 (7) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 2 (2) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 7 (7) | 6 (7) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 13 (15) | 17 (18) | 8 (9)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT02713204/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT02713204/SAP_001.pdf